CLINICAL TRIAL: NCT01061463
Title: Study of the Occupational Risk of Radiation-induced Cataracts Among Cardiologists
Brief Title: Occupational Cataracts and Lens Opacities in Interventional Cardiology : the O'CLOC Study
Status: Completed | Type: Observational
Sponsor: Sophie JACOB (Other Government)
Responsible Party: Sponsor-Investigator, Sophie JACOB, PhD, Institut de Radioprotection et de Surete Nucleaire
Organization: Institut de Radioprotection et de Surete Nucleaire (Other Government)
Other Study IDs: IRSN-09079
Record Dates: First submitted 2010-02-02; First posted 2010-02-03 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-04

CONDITIONS: Cataracts; Lens Opacities
Keywords: Radiation cataracts; Lens opacities; X-rays; Interventional Cardiologists; Electrophysiologists
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Exposed group: French coronary interventional cardiologists and cardiologists specializing in cardiac arrhythmias treatments (electrophysiologists), occupationally exposed to X-Rays
- Unexposed group: French non-interventional cardiologists and non medical workers, not occupationally exposed to X-Rays

SUMMARY:
The purpose of this study is to test the existence of an increased risk of cataracts among interventional cardiologists as compared to cardiologists not exposed to X-rays.

DETAILED DESCRIPTION:
This cross-sectional study includes cardiologists aged > 40 years: a group of interventional cardiologists (coronary interventionists and electrophysiologists) and a group of unexposed workers (including cardiologists). Individual information, including risk factors of cataracts (age, diabetes, myopia, etc. ...), are collected during a telephone interview. For the exposed group, a specific section of the questionnaire is focused on the occupational history, the description of the procedures (type, frequency, radiation protection tool) and will be used for the classification into "comparable exposure level" groups according to estimates of cumulative dose. For all participants, eye examinations are performed to specifically detect cataracts even in the early stages (lens opacities, LOCS III according to the international standard classification).

ELIGIBILITY:
Inclusion Criteria:

* aged at least 40 yrs old
* for interventional cardiologists: cumulated number of procedures > 2000

Exclusion Criteria:

* previous history of medical radiation exposure for radiotherapy or brain scans
* for non-interventional cardiologists: occupational history of interventional cardiologist

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Interventional and non-interventional cardiologists from public and private French hospitals/facilities, both groups of cardiologists being matched for age and gender.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2009-10; Primary Completion 2011-01 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Lens opacities | up to 1.5 year

SECONDARY OUTCOMES:
Visual acuity | up to 1.5 year
Major eye disorders (glaucoma, etc…) | up to 1.5 year

CONTACTS AND LOCATIONS:
Overall Officials: Sophie JACOB, PhD., Principal Investigator — Institut de Radioprotection et de Surete Nucleaire
Locations (1):
- IRSN, Fontenay-aux-Roses, France

REFERENCES:
- [Derived] Jacob S, Michel M, Spaulding C, Boveda S, Bar O, Brezin AP, Streho M, Maccia C, Scanff P, Laurier D, Bernier MO. Occupational cataracts and lens opacities in interventional cardiology (O'CLOC study): are X-Rays involved? Radiation-induced cataracts and lens opacities. BMC Public Health. 2010 Sep 8;10:537. doi: 10.1186/1471-2458-10-537. PMID 20825640